CLINICAL TRIAL: NCT05474755
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study on the Safety and Efficacy of GP681 Tablets in the Treatment of Acute Uncomplicated Influenza
Brief Title: To Assess the Efficacy of GP681 Tablet Versus Placebo in Patients With Acute Uncomplicated Influenza Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GP681-202201
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP681 40mg (Experimental): Patients in the GP681 40mg group will receive a single oral dose of GP681 tablet 40mg with 240mL water.
  Interventions: Drug: GP681 40mg
- placebo group (Placebo Comparator): Patients in the Placebo group will receive a single oral dose of GP681 Simulant 40mg with 240mL water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GP681 40mg — 2X20mg tablets taken orally
  Arms: GP681 40mg
Drug: Placebo — Placebo tablets matching GP681 40mg
  Arms: placebo group

SUMMARY:
This study will evaluate the efficacy, safety, and population pharmacokinetics of a single, oral dose of GP681 compared with placebo in patients aged 12 to 65 years with acute uncomplicated influenza virus infection

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged≥5 to≤65 years at the time of signing the informed consent form.
2. Patients with a diagnosis of influenza confirmed by all of the following:

   * Positive Influenza rapid antigen test or Polymerase chain reaction (PCR), and;
   * Fever (axillary temperature ≥37.3℃) in the predose examinations or > 4 hours after dosing of antipyretics if they were taken,and;
   * At least one of the following systemic symptoms and respiratory symptoms respectively associated with influenza are present with a severity of moderate or greater:

     1. Systemic symptoms: headache, fever or chills, muscle or joint aches, fatigue;
     2. Respiratory system symptoms: cough, sore throat, nasal congestion.
3. The time interval between the onset of symptoms and random enrollment is 48 hours or less. The onset of symptoms is defined as either:

   1. Time of the first increase in body temperature (axillary temperature ≥37.3℃)
   2. Time when the patient experiences at least one systemic or respiratory symptom related to influenza
4. Subjects of child-bearing potential who agree to use a highly effective method of contraception for 1 month after drug withdrawal.
5. Subjects and/or their guardian who are willing to provide written informed consent and consent to participate in the study, able to understand the study and comply with all study procedures, including patient health diary records.

Exclusion Criteria:

1. History of allergic reactions attributed to GP681 or any of the ingredients of its formulation.
2. Patients with influenza virus infection requiring inpatient treatment;
3. Known history of dysphagia or any gastrointestinal disease that affects drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, stomach after subtotal resection, etc.).
4. Treatment with anti-influenza virus drugs (oseltamivir, zanamivir, peramivir, favipiravir, arbidol, baloxavir marboxil, amantadine, or rimantadine) within 2 weeks before screening, or immunization with influenza vaccine within 6 months prior to enrollment;
5. Investigator suspects or confirms that patients with bronchitis, pneumonia, pleural effusion or interstitial disease through chest imaging examination.
6. Acute respiratory infection, otitis media or sinusitis within 2 weeks prior to Screening.
7. Patients with concurrent bacterial or (non-influenza) infections requiring systemic antimicrobial and/or antiviral therapy at the pre-dose examinations.
8. Positive nucleic acid test for COVID-19 in screening period.
9. Patients with severe or uncontrollable underlying diseases, including blood disorders, severe chronic obstructive pulmonary disease(COPD), liver disorders, kidney disorders, chronic congestive heart failure(NYHA III-IV), mental disorders;
10. Immunodeficiency,including malignant tumor, organ or marrow transplant, human immunodeficiency virus [HIV] infection, or patients receiving immunosuppressant therapy 3 months prior to enrollment.
11. Concomitant therapy with aspirin or salicylic acid.
12. Morbid obesity (Body mass index [BMI]≥30kg/m2)
13. Women who are pregnant, breastfeeding, or have a positive pregnancy test at the predose examinations. The following female patients who have documentation of either a or b below do not need to undergo a pregnancy test at the predose examinations:

    1. Postmenopausal women (defined as cessation of regular menstrual periods for 2 years or more and aged more than 50 years old)
    2. Women who are surgically sterile by hysterectomy, bilateral oophorectomy, or tubal ligation
14. Known history of alcohol abuse (Average weekly intake of alcohol is more than 14 units alcohol (1 units ≈ 360 mL beer, or 45 mL spirits with 40% content, or 150 mL wine) or drug abuse at screening;
15. Patients weighing <20 kg.
16. Has received any investigational agents or devices for any indication within 30 days prior to Screening.
17. Patients who, in the opinion of the Investigator, may not be qualified or suitable for the study.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of influenza symptoms | Up to Day 15
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Defined as the time from the start of treatment until the patient's body temperature returns to normal and all 7 flu symptoms (cough, sore throat, headache, nasal congestion, fever or chills, muscle or joint pain, fatigue) have alleviated (scoring 0 or 1 point) for at least 21.5 hours.

SECONDARY OUTCOMES:
Time to Cessation of Viral Shedding Determined by Virus Titer | Up to Day7
  Defined as the time between the initiation of the study treatment and first time when the virus titer was below the limit of detection.
Percentage of Participants With Positive Influenza Virus RNA by RT-PCR at Each Time Point | Days 2, 3, 5,7
  The percentage of patients positive for virus RNA by RT-PCR.
Percentage of Participants With Positive Influenza Virus Titer at Each Time Point | Days 2, 3, 5,7
  Virus titer was quantified from nasopharyngeal swabs by tissue culture methods.
Area Under the Concentration (AUC) of virus RNA by RT-PCR and AUC of virus titer | Up to Day 7
  AUC of the viral load by RT-PCR and AUC of viral titer measured from baseline to Day 7
Change From Baseline in Virus RNA (RT-PCR) at Each Time Point | Days 2, 3, 5,7
  Nasopharyngeal swabs were obtained for viral quantitation.
Change in the total score of 7 influenza symptoms | Up to Day15
  The composite symptom score is the total score of the 7 influenza symptoms(Sum of symptom scores) as assessed by the participant, and ranges from 0 to 21.
Time to alleviation of each influenza symptom | Up to Day15
  Defined as the time from the start of treatment to the start of the time period when the individual symptom was assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
Time to Alleviation of the Four Systemic Symptoms in Participants | Up to Day15
  Defined as the time between the initiation of the study treatment to the time when all 4 systemic symptoms (headache, fever or chills, muscle or joint pain, and fatigue) were assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
Time to Alleviation of the Three Respiratory Symptoms in Participants | Up to Day15
  Defined as the time from the start of study treatment to the time when all 3 respiratory symptoms (cough, sore throat and nasal congestion) were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours
Percentage of Participants Reporting Normal Temperature at Each Time Point | 12, 24, 48, 72, 96,120, 144 and168 hours after the initial dose of study treatment
  Defined as the percentage of patients whose axillary temperature dropped to less than 37.3 degree Celsius [ºC] after the initiation of study treatment
Time to Resolution of Fever | Up to Day15
  Defined as the time between the initiation of the study treatment and the resolution of fever. The resolution of fever was defined as the time when the participant's self-measured axillary temperature became less than 37.3ºC and was maintained at less than 37.3ºC for a duration of at least 21.5 hours.
Incidence of Influenza-related Complications | Up to Day15
  Defined as the percentage of subjects in the analysis population who experience each influenza-related complication (hospitalization, death, sinusitis, bronchitis, otitis media, and pneumonia) as an adverse event after the initiation of the study treatment.
Proportion of Patients and Frequency in Combination Use of Acetaminophen | Up to Day15
  The proportion of patients who use acetaminophen in the duration of the study.
Time to Return to Normal Activities of Daily Life | Up to Day15
  Defined as the time between the initiation of the study treatment and the return to normal activities of daily life. The return to normal activities of daily life is defined as the time when the subject assesses his/her activities as 10. Subjects with a baseline self-rated daily activity score of 10 are not included in this analysis.
Change from baseline in health-related quality of life according to EuroQol 5 dimensions 5 (EQ-5D-5L) questionnaire | Up to Day15
  The EQ-5D-5L is a self-reported health status questionnaire that consists of six questions used to calculate a health utility score for use in health economic analysis. There are two components to the EQ-5D-5L: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, phd, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- The First People's Hospital of Wenling, Wenling, Zhejiang, China

REFERENCES:
- [Derived] Wang Y, Wang H, Zhang Y, Ma A, Liu D, Li X, Yang G, Deng M, Wang S, Liu Y, Liu C, Ge F, Wang S, Yu Y, Feng G, Xiao Z, Li X, Sun Y, Chen X, Cao Z, Ding Y, Wu X, Wei J, Cao B. Single-dose suraxavir marboxil for acute uncomplicated influenza in adults and adolescents: a multicenter, randomized, double-blind, placebo-controlled phase 3 trial. Nat Med. 2025 Feb;31(2):639-646. doi: 10.1038/s41591-024-03419-3. Epub 2025 Jan 7. PMID 39775042